CLINICAL TRIAL: NCT05499767
Title: HEPPI: A Randomized Controlled Trial of the Efficacy of a Cognitive-Emotional Intervention for Homebound Older Adults
Brief Title: HEPPI: Efficacy of a Cognitive-Emotional Intervention for Homebound Older Adults
Acronym: HEPPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Andreia Jesus, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HEPPIEfficacy/CINEICC; SFRH/BD/146170/2019 (Other Grant/Funding Number: Foundation for Science and Technology (FCT))
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Depressive Symptoms; Anxiety State
Keywords: Homebound Older Adults; Mild Cognitive Impairment; Depressive and Anxious Symptomatology; Cognitive-Emotional Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEPPI (Experimental): The HEPPI group attends weekly 90-minute intervention sessions at the participants' homes.
  Interventions: Behavioral: HEPPI
- Treatment as Usual (TAU) (No Intervention): The TAU group receives access to HEPPI at the end of the study.

INTERVENTIONS:
Behavioral: HEPPI — Homebound Elderly People Psychotherapeutic Intervention
  Arms: HEPPI

SUMMARY:
The main goal of this research is to assess the efficacy of a 10-week home-delivered cognitive-emotional intervention program for homebound older adults presenting Mild Cognitive Impairment (MCI) and depressive and/or anxiety symptoms. The Homebound Elderly People Psychotherapeutic Intervention (HEPPI) combines cognitive training, psychotherapeutic techniques, and compensatory strategy training, and was designed to optimize memory function and to reduce depressive or anxious symptomatology of these older adults.

A two-arm randomized controlled trial (RCT) is conducted to investigate the efficacy of the HEPPI among the homebound older population.

DETAILED DESCRIPTION:
The present study aims to assess the efficacy of a cognitive-emotional intervention (the HEPPI program) for homebound older adults with MCI and depressive and/or anxious symptomatology.

The research design of the trial followed the methodological recommendations for conducting goropsychoterapy research. Moreover, a pilot RCT was conducted prior to the present RCT, in order to assess the feasibility, acceptability, and preliminary efficacy of the HEPPI. Appropriate adjustments to the HEPPI protocol were carried out considering the results.

The present study is a two-arm RCT comparing the intervention condition (HEPPI) to a treatment as usual (TAU) control group. The sample includes community-dwelling older adults who do not leave home more often than once a week. Homebound older adults are recruited from the community through contact with their health care networks. A minimum number of 79 participants per condition will be required (N=158). Accounting for an expected 20% attrition rate, an anticipated sample of 198 participants will be enrolled in the study. Participants who demonstrate interest in the study are informed of the goals and procedures of the research and asked to provide informed consent before eligibility assessment. Eligible participants are randomly assigned to the HEPPI or the TAU group.

Homebound older adults are asked to complete baseline, post-intervention, and 3-month follow-up assessments. Assessments include neuropsychological tests to assess cognition function, psychological health, subjective memory complaints, quality of life, functional status, perceived loneliness, and personality. The study procedures take place at the participants' homes.

ELIGIBILITY:
Inclusion Criteria:

* Homebound older adults aged 65 years and older;
* MoCA score 1 to 1.5 standard deviation below the mean for age- and education- adjusted norms;
* FCSRT total immediate and delayed recall scores ≤ 35 and ≤ 12, respectively;
* Presence of subjective memory complaints (SMCS score ≥ 3);
* Presence of depressive symptomatology (GDS-30 score ≥ 11);
* Presence of anxious symptomatology (GAI score ≥ 8);
* No significant impact from cognitive impairment on daily functional capacity;
* Residence in mainland Portugal;

Exclusion Criteria:

* Presence or history of significant neurological conditions;
* Presence of severe psychiatric illnesses;
* Presence of comorbid medical conditions associated with cognition decline;
* Use of psychotropic medication for less than three months;
* Presence of alcoholism or toxicomania;
* Significant impairment of vision, hearing, communication, or manual dexterity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in Episodic Memory | Baseline, post-intervention, and 3-month follow-up
  Logical Memory of the Wechsler Memory Scale-III (LM) | Higher scores indicate a better outcome
Changes in Depressive Symptomatology | Baseline, post-intervention, and 3-month follow-up
  Measured by Geriatric Depression Scale-30 (GDS-30) | Lower scores indicate a better outcome
Changes in Anxious Symptomatology | Baseline, post-intervention, and 3-month follow-up
  Measured by Geriatric Anxiety Inventory (GAI) | Lower scores indicate a better outcome

SECONDARY OUTCOMES:
Changes in General Cognitive Function | Baseline, post-intervention, and 3-month follow-up
  Measured by Addenbrooke's Cognitive Examination-Revised (ACE-R) | Higher scores indicate a better outcome
Changes in Attentional Control | Baseline, post-intervention, and 3-month follow-up
  Measured by Digit Symbol-Coding of the Wechsler Adult Intelligence Scale-III (DSC) | Higher scores indicate a better outcome
Changes in Subjective Memory Complaints | Baseline, post-intervention, and 3-month follow-up
  Measured by Subjective Memory Complaints Scale (SMCS) | Lower scores indicate a better outcome
Changes in Perceived Quality of Life | Baseline, post-intervention, and 3-month follow-up
  Measured by European Portuguese World Health Organization Quality of Life-Old Module (WHOQOL-OLD) | Higher scores indicate a better outcome
Changes in Functional Status | Baseline, post-intervention, and 3-month follow-up
  Measured by Adults and Older Adults Functional Assessment Inventory (IAFAI) | Lower scores indicate a better outcome
Changes in Loneliness | Baseline, post-intervention, and 3-month follow-up
  Measured by UCLA Loneliness Scale (UCLA) | Lower scores indicate a better outcome

OTHER OUTCOMES:
Personality Traits | Baseline
  Measured by NEO Five-Factor Inventory (NEO-FFI)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive Behavioral Intervention (CINEICC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jesus AG, de Lima MP, Vilar M, Pachana NA. Homebound elderly people psychotherapeutic intervention (HEPPI): Exploring the mediating role of loneliness. Arch Gerontol Geriatr. 2024 Mar;118:105308. doi: 10.1016/j.archger.2023.105308. Epub 2023 Dec 3. PMID 38101250
- [Derived] Jesus AG, Lima MP, Vilar M, Pachana NA. HEPPI: a randomized controlled trial of the efficacy of a cognitive-emotional intervention for homebound older adults. Aging Ment Health. 2024 Mar-Apr;28(3):491-501. doi: 10.1080/13607863.2023.2260760. Epub 2023 Sep 25. PMID 37747057